CLINICAL TRIAL: NCT02771639
Title: Early Periprosthetic Joint Infection and Debridement, Antibiotics and Implant Retention in Arthroplasty for Femoral Neck Fracture
Brief Title: Early Periprosthetic Joint Infection and Outcome Debridement, Antibiotics and Implant Retention
Acronym: DAIR
Status: Completed | Type: Observational
Sponsor: Sundsvall Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DAIR_SM
Record Dates: First submitted 2016-05-08; First posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Femoral Neck Fracture; Infection
Keywords: Hip arthroplasty; periprosthetic joint infection; outcome
MeSH Terms: conditions — Femoral Neck Fractures; Infections | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Femoral neck fractures: Patients admitted to Sundsvall hospital for a displaced femoral neck fracture and treated with a hip arthroplasty
  Interventions: Procedure: Hip arthroplasty

INTERVENTIONS:
Procedure: Hip arthroplasty — Treatment with a hip arthroplasty (semi- or total hip arthroplasty) for a displaced femoral neck fracture

SUMMARY:
Introduction Periprosthetic joint infection (PJI) is a severe complication to hip arthroplasty for femoral neck fractures (FNF). Debridement, antibiotics and implant retention (DAIR) is recommended in early PJI in association with stable implants. Few studies have evaluated the outcome of DAIR in this fragile population.The purpose of this study was to analyze risk factors for PJI and the short-term outcome of DAIR in FNF patients treated with a hip arthroplasty.

Methods A consecutive series of patients had been treated with either a total hip arthroplasty or a hemi hip arthroplasty for a displaced FNF at our institution. Data were retrospective analysed.

ELIGIBILITY:
Inclusion Criteria:

* Displaced femoral neck fracture
* Treated with a primary hip arthroplasty

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with a hip arthroplasty for a displaced femoral neck fracture at Sundsvall hospital, Sweden between 2006 and 2015. All patients were included.
Sampling Method: Non-Probability Sample
Enrollment: 736 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Rate of periprosthetic joint infection | 1 year
  The incidence of periprosthetic joint infection

SECONDARY OUTCOMES:
The rate of healed periprosthetic joint infections after treatment with surgical debridement. | 6 months
  The rate of healed periprosthetic joint infections after treatment with surgical debridement.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Mukka, M.D, Ph.D, Principal Investigator — Umeå University

IPD SHARING:
Plan to Share IPD: Undecided
No individual data

REFERENCES:
- [Background] Osmon DR, Berbari EF, Berendt AR, Lew D, Zimmerli W, Steckelberg JM, Rao N, Hanssen A, Wilson WR; Infectious Diseases Society of America. Executive summary: diagnosis and management of prosthetic joint infection: clinical practice guidelines by the Infectious Diseases Society of America. Clin Infect Dis. 2013 Jan;56(1):1-10. doi: 10.1093/cid/cis966. PMID 23230301
- [Background] Dale H, Fenstad AM, Hallan G, Havelin LI, Furnes O, Overgaard S, Pedersen AB, Karrholm J, Garellick G, Pulkkinen P, Eskelinen A, Makela K, Engesaeter LB. Increasing risk of prosthetic joint infection after total hip arthroplasty. Acta Orthop. 2012 Oct;83(5):449-58. doi: 10.3109/17453674.2012.733918. PMID 23083433
- [Background] Edwards C, Counsell A, Boulton C, Moran CG. Early infection after hip fracture surgery: risk factors, costs and outcome. J Bone Joint Surg Br. 2008 Jun;90(6):770-7. doi: 10.1302/0301-620X.90B6.20194. PMID 18539671
- [Background] Fisman DN, Reilly DT, Karchmer AW, Goldie SJ. Clinical effectiveness and cost-effectiveness of 2 management strategies for infected total hip arthroplasty in the elderly. Clin Infect Dis. 2001 Feb 1;32(3):419-30. doi: 10.1086/318502. Epub 2001 Jan 26. PMID 11170950
- [Background] Noailles T, Brulefert K, Chalopin A, Longis PM, Gouin F. What are the risk factors for post-operative infection after hip hemiarthroplasty? Systematic review of literature. Int Orthop. 2016 Sep;40(9):1843-8. doi: 10.1007/s00264-015-3033-y. Epub 2015 Nov 27. PMID 26611729